CLINICAL TRIAL: NCT02111005
Title: Influence of Smoking on Fibroblast Apoptosis in Patients With Chronic and Aggressive Periodontitis
Brief Title: Smoking Influence on Apoptosis in Periodontitis
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-Perio-01-2014
Record Dates: First submitted 2014-03-14; First posted 2014-04-10 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Periodontitis; Aggressive Periodontitis
Keywords: apoptosis; periodontal disease; smoking
MeSH Terms: conditions — Chronic Periodontitis; Aggressive Periodontitis; Periodontal Diseases; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Smoking Aggressive Periodontitis group: This group comprises 20 patients who are smokers and aged < 35 years and diagnosed with rapid attachment loss with periodontal pocket depth (PD) > 4 mm around at least three teeth other than the first molars and incisors. Rapid bone destruction (>50%bone loss at diseased sites). Weak relationship between dental plaque and the severity of gingival inflammation.
- Smoking Chronic Periodontitis group: This group comprises 20 patients who are smokers and aged > 45 years and have presence of ≥2 non-adjacent sites per quadrant that were not first molars or incisors, with probing depth (PD) ≥5 mm, which bleed on gentle probing. The demonstrated radiographic bone loss ≥30% of the root length, patient with poor oral hygiene, the amount of accumulated plaque commensurate with the amount of clinical attachment level (CAL)
- Non-smoking Aggressive Periodontitis grp: This group comprises 20 patients who are age- and sex- matched to the 'Smoking Aggressive Periodontitis group' and are non-smokers suffering from aggressive periodontitis.
- Non-smoking Chronic periodontitis grp: This group comprises 20 patients who are age- and sex-matched to the 'Smoking Chronic Periodontitis group' and are non-smokers suffering from chronic periodontitis.

SUMMARY:
Apoptosis is an evolutionary form of physiological cell death. Studies suggest that apoptosis is involved in the pathogenesis of periodontal diseases. Human gingival fibroblasts (HGF) have an important role in the periodontal immune response. It is believed that HGF can be diminished and/or eliminated by means of apoptosis.

Smoking is one of the most common risk factor of periodontal disease. Studies indicated that smoking can increase the risk of periodontitis by enhancing the apoptosis of gingival fibroblast.

The purpose of this study is to determine and to investigate apoptosis of HGF in gingival biopsies collected from smokers and non smokers who are diagnosed with chronic periodontitis or aggressive periodontitis.

Eighty subjects will be invited to participate in this study. Patients will be allocated into four groups (20 patients each). Gingival biopsies will be obtained from the base of papillae during surgical treatment (open flap curettage) and will be examined by Immuno-histochemical analysis. Immune-staining will be done using p53 monoclonal mouse anti-human antibody.

DETAILED DESCRIPTION:
Background:

The mechanisms responsible for gingival tissue damage are poorly understood, and both immune-mediated reactions and direct cytopathic effects of bacteria maybe involved. Based on direct effect of bacteria in cell cultures, it has been suggested that apoptosis might play an important role in periodontitis (Chen 1994).

Programmed cell death (apoptosis) is normal physiologic process that contributes to maintaining tissue homeostasis. The process of apoptosis can be modulated by various stimuli hormones, cytokines, growth factors, infections and immune-responses (Renehan et al. 2001).

Among other factors, the products of two genes that encode protein p53 and Bcl-2 have been shown to play fundamental regulatory role in apoptosis. P53 is the protein product of tumor-suppressor gene, and expression of P53 can induce apoptosis. This protein is also implicated in the regulation of tissue dynamics, and is specifically thought to induce apoptosis in terminally differentiated cells, including inflammatory cells (Bulut et al.2006).

Fibroblast is a type of cell that synthesizes the extracellular and collagen in connective tissue. It plays a critical role in wound healing. Fibroblasts are the most common cells in connective tissue. The main function of fibroblasts is to maintain the structural integrity of connective tissue by continuously secreting precursors of extracellular matrix. it was reported that apoptosis levels increased in gingivitis and periodontitis (Jarenberg et al. 2002).

Cigarette smoking is a risk factor for many diseases, and recent evidence indicates that smoking adversely influences periodontal health. A number of epidemiologic studies have shown strong association between smoking and prevalence and severity of periodontitis (Bostrom et al. 1998). Whereas, the pathogenesis of periodontitis in smokers is poorly understood there are data suggesting that smoking effects on the periodontal tissues include defects in neutrophil function, impaired serum antibody responses to periodontal pathogens, and potentially diminished gingival fibroblast function (Shivanaikar et al. 2001). Smokers are considered a high-risk group for periodontitis, and smoking history is a useful clinical predictor of future disease activity (Hanokia et al. 2000).

Aims of the study:

* Investigation of the effects of smoking on fibroblasts apoptosis in smokers with periodontitis compared to non-smokers with periodontitis using immuno-histochemical methods.
* Comparison of apoptosis levels of gingival fibroblasts between chronic and aggressive periodontitis.

Materials and methods:

A total of 80 subjects will be invited to participate in this study from the patients referred to the Department of Periodontology, Faculty of Dentistry, University of Damascus. The study will be approved by a specific Review Board. Subjects will be recruited according to specific inclusion criteria after completion of medical and dental history questionnaires. Patients will sign a consent form after being advised about the nature of the study.

The selection of patients will be made according of the criteria approved by the 1999 international world workshop for a classification system of periodontal diseases and conditions (Armitage 1999) using five clinical parameters and full mouth or panoramic radiographs for diagnosis.

Subjects will be allocated into four groups:

* Smoking Chronic Periodontitis group (ChP-S): comprise 20 patients who are smokers and aged > 45 years and have presence of ≥2 non-adjacent sites per quadrant that were not first molars or incisors, with probing depth (PD) ≥5 mm, which bleed on gentle probing. The demonstrated radiographic bone loss ≥30% of the root length, patient with poor oral hygiene, the amount of accumulated plaque commensurate with the amount of clinical attachment level (CAL)
* Non-smoking Chronic periodontitis group (ChP-NS): comprise 20 age-sex matched patients who are non-smokers and have chronic periodontitis.
* Smoking Aggressive Periodontitis group (AgP-S): comprise 20 patients who are smokers and aged < 35 years and diagnosed with rapid attachment loss with periodontal pocket depth (PD) > 4 mm around at least three teeth other than the first molars and incisors. Rapid bone destruction (>50%bone loss at diseased sites). Weak relationship between dental plaque and the severity of gingival inflammation.
* Non-smoking Aggressive periodontitis group (AgP-NS): comprise 20 age- and sex matched patients who are non-smokers and have aggressive periodontitis.

Clinical measurements:

A standard periodontal probe will be used for recording periodontal indices at six sites per tooth. The examined clinical parameters include bleeding on probing (BOP), plaque index (PI), clinical attachment loss (CAL) and periodontal pocket depth (PPD) and gingival index (GI).

Biopsy collection and analysis

* The biopsy samples will be obtained from patients during surgical treatment (open flap curettage) where biopsy is taken from the base area of papilla.
* Samples will be placed in 10% formalin.
* The samples will be then installed in paraffin wax.
* Samples will be analyzed in the by means of p53 monoclonal mouse anti-human antibody.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Syrian descent
* Systemically healthy
* Have at least 20 teeth

Exclusion criteria:

* Periodontal treatment during the last three months
* History of major systemic diseases
* Consumption of antibiotics or anti-inflammatory drugs in the last three months
* Smoking
* Alcohol consumption
* Pregnant and lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 80 subjects will be invited to participate in this study from the patients referred to the Department of Periodontology, Faculty of Dentistry, University of Damascus. Patients should have a diagnosis of periodontitis (either chronic or aggressive). Any candidate will be approached and informed about this clinical study with the relevant information sheet. Informed consent forms will be obtained.Using five clinical parameters and full mouth or panoramic radiographs, the participants will be allocated to four groups according to their condition as well as their smoking habit. The description of these groups has given before.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
P53 levels in gingival biopsy samples | The measurement will be performed at T0 (baseline measurement) once the sample has been recruited
  This variable is going to be measured by an immunohistochemical analysis

SECONDARY OUTCOMES:
presence or absence of fibroblasts' apoptosis in the gingival tissues | The measurement will be performed at T0 (baseline measurement) once the sample has been recruited
  this variable is going to be measured by an immunohistochemical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ali Abou Sulaiman, DDS MSc PhD, Principal Investigator — University of Damascus Dental School, Department of Periodontology; Sharif Barakat, DDS MSc Phd, Study Director — University of Damascus Dental School, Department of Periodontology
Locations (2):
- Syria (2):
  - Department of Periodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate
  - Ali Abou Sulaiman, Damascus, Syrian Arab Republic

REFERENCES:
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Bostrom L, Linder LE, Bergstrom J. Clinical expression of TNF-alpha in smoking-associated periodontal disease. J Clin Periodontol. 1998 Oct;25(10):767-73. doi: 10.1111/j.1600-051x.1998.tb02368.x. PMID 9797047
- [Background] Bulut S, Uslu H, Ozdemir BH, Bulut OE. Expression of caspase-3, p53 and Bcl-2 in generalized aggressive periodontitis. Head Face Med. 2006 Jun 20;2:17. doi: 10.1186/1746-160X-2-17. PMID 16787530
- [Background] Chen Y, Zychlinsky A. Apoptosis induced by bacterial pathogens. Microb Pathog. 1994 Oct;17(4):203-12. doi: 10.1006/mpat.1994.1066. PMID 7715420
- [Background] Jarnbring F, Somogyi E, Dalton J, Gustafsson A, Klinge B. Quantitative assessment of apoptotic and proliferative gingival keratinocytes in oral and sulcular epithelium in patients with gingivitis and periodontitis. J Clin Periodontol. 2002 Dec;29(12):1065-71. doi: 10.1034/j.1600-051x.2002.291203.x. PMID 12492905
- [Background] Hanioka T, Tanaka M, Ojima M, Takaya K, Matsumori Y, Shizukuishi S. Oxygen sufficiency in the gingiva of smokers and non-smokers with periodontal disease. J Periodontol. 2000 Dec;71(12):1846-51. doi: 10.1902/jop.2000.71.12.1846. PMID 11156041
- [Background] Renehan AG, Booth C, Potten CS. What is apoptosis, and why is it important? BMJ. 2001 Jun 23;322(7301):1536-8. doi: 10.1136/bmj.322.7301.1536. No abstract available. PMID 11420279
- [Background] Shivanaikar S, Faizuddin M and Bhatt K. Influence of smoking on fibroblast apoptosis in chronic periodontitis. RGUHS J Dent Sciences. 2001; 3: 9-14